CLINICAL TRIAL: NCT03108417
Title: Home Study of Subjects With Obstructive Sleep Apnea Who Have Previously Completed an In-Lab Continuous Negative External Pressure (cNEP) Titration and Were Considered to be "Responders"
Brief Title: Home Study of Subjects Who Have Completed a Previous Continuous Negative External Pressure (cNEP) Clinical Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no eligible subjects were available for recruitment
Sponsor: Sommetrics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOM-013
Record Dates: First submitted 2017-03-25; First posted 2017-04-11 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- cNEP (Experimental): continuous negative external pressure will be used nightly by all participants
  Interventions: Device: continuous negative external pressure

INTERVENTIONS:
Device: continuous negative external pressure — continuous negative external pressure will be applied to the anterior neck at night
  Other Names: cNEP

SUMMARY:
This study is designed to determine whether subjects who were responders to cNEP during an overnight sleep lab titration in a previous clinical trial, Study SOM-012, will maintain a response throughout the night for up to two weeks in a home setting. It will also be determined whether two weeks of home use of cNEP is associated with any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* must have completed study SOM-012 and been categorized as a "responder"
* the subject agrees to participation by signing an informed consent statement

Exclusion Criteria:

* medical or social circumstances have changed since participation in SOM-012 such that continued use of cNEP may provide questionable benefit or associated with increased risk

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Reduction in baseline apnea hypopnea index from baseline | End of Week 2 of home use
  Reduction in apnea hypopnea index (AHI) from the baseline value of >50% and also <15/hr

SECONDARY OUTCOMES:
Collection of adverse events | two week study period
  Collection of adverse events
Apnea hypopnea index, as measured by home sleep testing | two weeks
  Comparison of AHI from home sleep testing in this study to those of the polysomnogram (PSG) in SOM-012

OTHER OUTCOMES:
Clinical global impression of cNEP experience | end of week two of home use
  Assessment of the tolerability of cNEP to the subject via a clinical global impression scale
Bed partner's views of cNEP via a clinical global impression scale | end of two weeks of home use
  Determination of the bed partner's views of the subject using cNEP in the home setting using a clinical global impression scale

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Kram, MD, Principal Investigator — California Center for Sleep Disorders
Locations (1):
- California Center for Sleep Disorders, Alameda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided